CLINICAL TRIAL: NCT02140411
Title: Chilean Interventional Open Label Pilot Study, to Assess the Efficacy and Safety of Lucentis® (Ranibizumab Intravitreal Injections) in Patients With Visual Impairment Due to Diabetic Macular Edema.
Brief Title: Efficacy and Safety of Lucentis® (Ranibizumab Intravitreal Injections) in Chilean Patients With Diabetic Macular Edema.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DCL01
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2018-10

CONDITIONS: Retinal Vein Occlusion; Age Related Macular Degeneration
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ranibizumab (Experimental): Ranibizumab treatment
  Interventions: Drug: Ranibizumab Intravitreal injections

INTERVENTIONS:
Drug: Ranibizumab Intravitreal injections — Ranibizumab intravitreal injections 3 months 1 per month and after PRN treatment.

SUMMARY:
Ranibizumab is a humanized anti-vascular endothelial growth factor (VEGF) monoclonal antibody fragment approved in Chile by the Instituto de Salud Pública for the treatment of diabetic macular edema (DME), retinal vein occlusion and age-related macular degeneration.

Currently, there is limited epidemiologic information in Chile regarding the incidence of DME and limited experience of anti-VEGF hospital therapy. This study will evaluate the efficacy of intravitreal ranibizumab in Chilean DME patients, to investigate the anatomical and functional improvement following this treatment and to increase the local experience regarding the use of anti-VEGF in the treatment of diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of macular edema due to diabetes (confirmed by fundus photography, and/or fluorescein angiography, and/or OCT) in at least one eye.
2. Vision impairment due to DME (BCVA ETDRS letter score at 4 meters between 20 and 70 letters (6/12 - 3/60 at Snellen chart).

Exclusion Criteria:

1. Laser photocoagulation in the study eye for the last 3 months.
2. Any history of any intraocular surgery in the study eye within the past 3 months.
3. Blood pressure >160/100 mmHg.
4. Proliferative Diabetic Retinopathy.

Any other protocol inclusion/exclusion criteria that may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04-25 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Providencia, Santiago de Chile, Chile

REFERENCES:
- [Background] Wild S, Roglic G, Green A, Sicree R, King H. Global prevalence of diabetes: estimates for the year 2000 and projections for 2030. Diabetes Care. 2004 May;27(5):1047-53. doi: 10.2337/diacare.27.5.1047. PMID 15111519
- [Result] Ciulla TA, Amador AG, Zinman B. Diabetic retinopathy and diabetic macular edema: pathophysiology, screening, and novel therapies. Diabetes Care. 2003 Sep;26(9):2653-64. doi: 10.2337/diacare.26.9.2653. PMID 12941734

RESULTS

PARTICIPANT FLOW:
Groups:
- Ranibizumab: Ranibizumab 0.5 mg administered as an intravitreal injection
Period: Overall Study
Arm/Group | Ranibizumab
Started | 21
Completed | 20
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) include all patients who received at least one dose of study medication, and have at least one post-baseline efficacy assessment. The FAS is analyzed according to the intention to treat ideal.
Arm/Group | Ranibizumab
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.43 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Best Correct Visual Acuity (BCVA)
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (EDTRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. A positive change from baseline of BCVA indicates improvement.
Time Frame: baseline, week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 20
Letters | 9.55 (6.57)

2. Secondary Outcome: Change From Baseline in Best-corrected Visual Acuity (BCVA) After Week 4, 8, 12, 24 and 36
Description: BCVA was assessed in a sitting position using Early Treatment Diabetic Retinopathy Study (ETDRS)-like visual acuity (VA) testing charts at an initial testing distance of 4 meters. A positive change from baseline indicated improvement.
Time Frame: Baseline, Week 4, 8, 12, 24 and 36
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ranibizumab
Number analyzed (Participants) | 20
Letters
  Week 4 | 5.65 (5.25)
  Week 8 | 6.90 (4.27)
  Week 12 | 8.50 (6.13)
  Week 24 | 8.05 (7.32)
  Week 36 | 8.40 (7.18)

3. Secondary Outcome: Change Over Time of the Intraretinal Thickness in Optical Coherence Tomography (OCT)
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation, an increase in thickness as compared to baseline may indicate a progression of the underlying disease.
Time Frame: Baseline, week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Ranibizumab
Number analyzed (Participants) | 20
Microns
  Right eye | 388.50 (151.39)
  Left eye | 367.06 (91.44)

4. Secondary Outcome: Number of Participants Receiving Injections of Ranibizumab 0.5 mg Over a 48 Week Treatment Period.
Time Frame: Week 48
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 20
Count of participants | 7

5. Secondary Outcome: Number of Participants With Letters Gain / Loss at Week 52
Description: Number of participants with letters correctly identified were performed with the patient in a sitting position using ETDRS-like visual acuity testing charts at a testing distance of 4 meters.
Time Frame: Baseline, Week 52
Population: as for baseline characteristics
Measure: Number; unit: Count of Participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 21
Count of Participants
  5 or more letters gained | 14
  10 or more letters gained | 8
  15 or more letters gained | 5
  5 or more letters lost | 0
  10 or more letters lost | 0
  15 or more letters lost | 0

6. Secondary Outcome: Change in Mean Visual Function Questionnaire (VFQ-25)
Description: "Visual functioning was assessed by the patient using the National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25) on a scale from 0 to 100, where 0 = worst possible score and 100 = best. A positive change value indicates a perceived improvement in visual functioning, while a negative change value indicates a worsening."
Time Frame: Baseline, week 48
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ranibizumab
Number analyzed (Participants) | 20
Score on a scale
  General health | 12.50 (28.68)
  General vision | 13 (14.90)
  Ocular pain | 11.88 (23.81)
  Near activities | 7.50 (16.64)
  Distance activities | 9.62 (16.26)
  Social Functioning | 13.13 (15.95)
  Mental health | 9.69 (31.90)
  Role difficulties | 10.63 (34.24)
  Dependency | 13.75 (26.94)
  Driving | -0.0 (22.05)
  Color vision | 15 (27.39)
  Peripheral vision | 7.50 (31.52)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit, up to 14 months.
Description: AE additional description
Groups:
- Ranibizumab 0.5 mg: Ranibizumab 0.5 mg administered as an intravitreal injection
Arm/Group | Ranibizumab 0.5 mg
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=21)
Conjunctival haemorrhage (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Ischaemic stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=21)
Conjunctival haemorrhage (Eye disorders) | 2
Conjunctivitis allergic (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Ocular hypertension (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Influenza like illness (General disorders) | 1
Nodule (General disorders) | 1
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Intraocular pressure increased (Investigations) | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Migraine (Nervous system disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Menopause (Social circumstances) | 1
Carpal tunnel decompression (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety